CLINICAL TRIAL: NCT04755738
Title: Almonertinib Plus Microwave Ablation Versus Almonertinib in Previously Untreated，Advanced Non-small Cell Lung Cancer, a Randomized，Controlled，Phase II Clinical Trial
Brief Title: Almonertinib Plus Microwave Ablation in Advanced Non-small Cell Lung Cancer
Acronym: MWA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Lili Cao, Head of the department of oncology, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QianfoshanH O
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; microwave ablation; epidermal growth factor receptor; progression free survival; overall survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Almonertinib plus Microwave ablation group (Experimental): Patients in the group were treated with both targeted therapy and microwave ablation. Patients were treated with Almonertinib with the dose of 110mg once daily firstly. When the best response achieved, microwave ablation was conducted in the primary tumors, and then followed by Almonertinib treatments.
  Interventions: Combination Product: Almonertinib plus microwave ablation
- Almonertinib group (Active Comparator): Patients in the group were treated with Almonertinib with the dose of 110mg once daily until disease progression, death or intolerable adverse events.
  Interventions: Combination Product: Almonertinib plus microwave ablation

INTERVENTIONS:
Combination Product: Almonertinib plus microwave ablation — Patients were treated with almonertinib firstly.When almonertinib achieved the maximal response, microwave ablation was conducted on the primary lung tumors.
  Other Names: Microwave ablation

SUMMARY:
Almonertinib, as a third-generation EGFR-TKI, has been used for the treatment of advanced non small cell lung cancer. How to improve the progression free survival in advance was a challenge. Our previous study showed that first-line EGFR-TKIs plus microwave ablation had PFS survival advantage versus EGFR-TKIs alone. So we conducted this prospective study to verify the efficacy and safety of the combination in a randomized, controlled, phase II clinical trial.

DETAILED DESCRIPTION:
Almonertinib, as a third-generation EGFR-TKI, has been used for the treatment of advanced non small cell lung cancer. How to improve the progression free survival in advance was a challenge. Our previous study showed that first-line EGFR-TKIs plus microwave ablation had PFS survival advantage versus EGFR-TKIs alone. So we conducted this prospective study to verify the efficacy and safety of the combination in a randomized, controlled, phase II clinical trial. Patients were assigned into two groups.In the experiment group, patients were treated with both Almonertinib and microwave ablation. In the control group, patients were treated with Almonertinib alone. The primary end point was progression free survival. Second endpoints included overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically verified non-small-cell lung cancer;
2. Clinical stage of IIIB/IIIC/IV (including postoperative recurrence) ;
3. EGFR Exon 19del or Exon 21 L858R mutations;
4. No previous anti-tumor therapy including chemotherapy, radiotherapy or local thermal ablation (except adjuvant radiotherapy after lung cancer surgery) ;
5. ECOG PS 0-1;
6. Anticipated survival time ≥3 months;
7. At least one measurable lesions (according to RECIST 1.1, CT scan length ≥10mm, CT scan short diameter ≥15mm) except the ablation lesions (primary lesion or the largest recurrent lesion) ;
8. Asymptomatic brain metastasis;
9. The routine laboratory examination was normal (blood routine, liver and kidney function, blood coagulation function, etc The standard of blood routine examination should be met (No blood transfusion and blood products within 14 days) ; ANC≥1.5×109/L; PLT ≥80×109/L. B. Biochemical examination should meet the following criteria: TBIL≤ 1.5 ULN; ALT, Ast ≤ 2.5 ULN).
10. Adequate tissue specimens for further analysis.
11. Patients with potential fertility need to use a medically approved contraceptive method (such as intrauterine device, birth control pills or condoms) during and within 1 month after the end of the study period; The serum or urine HCG test must be negative within 72 hours before admission to the study, and must be non-lactation period; (12)18-80 years old;

(13)Patients signed informed consent;

Exclusion Criteria:

1. Mixed lung cancer including neuroendocrine or small-cell lung cancer;
2. Multiprimary tumors during the past 5 years;
3. Uncontrolled pleural or pericardial effusion;
4. Patients with a history of interstitial lung disease disease or moderate to severe diffuse dysfunction of the lung;
5. A severe infection (CTCAE > 2) during the past 4 weeks, such as severe pneumonia, bacteremia, infection complications, etc. requiring hospitalization;
6. baseline chest radiographic examination revealed active pulmonary inflammation.
7. The patients experienced acute cardiac cerebrovascular disease such as acute cerebral infarction and acute coronary syndrome within 1 month, (8) The cardiovascular clinical symptoms or diseases were not well controlled, including the following cases: There is local active Ulcer Focus, and stool occult blood {(+ +) can not be included in the group } ; within 2 months, there are black stool, hematemesis history;
8. Abnormal coagulation function with bleeding tendency;
9. Congenital or acquired immune deficiency (such as HIV infection) or active hepatitis (Hepatitis B reference: HBV DNA test above the normal limit; Hepatitis C reference: HCV virus or RNA test above the normal limit) ;
10. Patients with a history of psychotropic substance abuse who are unable to quit or who have a mental disorder;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From the date of randomization to the date of disease progression or death for any causes，whichever came first, assessed up to 36 months.
  progression free survival

SECONDARY OUTCOMES:
OS | From the date of randomization to the date of death, assessed up to 36 months.
  overall survival

OTHER OUTCOMES:
AE | From the date of randomization to the date of disease progression or death，whichever came first, assessed up to 36 months.
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Ye, Jinan, SD, China

IPD SHARING:
Plan to Share IPD: No
It depends.